CLINICAL TRIAL: NCT06593496
Title: Addressing Cardiometabolic Health In Populations Through Early Prevention in the Great Lakes Region Project 1 - Epidemiology (ACHIEVE P1-EPI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Phillip Levy, Professor, Assistant Vice President for Translational Sciences and Clinical Research Innovation, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Project-5757
Record Dates: First submitted 2024-07-30; First posted 2024-09-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Hypertension; High Blood Pressure
Keywords: Epidemiology; Mobile Health Unit; Prospective
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Text Message (Experimental): Participants assigned to the interventional group will receive a text message reminding them to take their blood pressure.
  Interventions: Behavioral: Text Message Reminder
- Control/No Text Message (No Intervention): Those assigned to the usual care group will not receive a reminder text message.

INTERVENTIONS:
Behavioral: Text Message Reminder — Randomized selection of recruited participants that will receive text messages reminding them to take their blood pressure.
  Arms: Text Message

SUMMARY:
This project is part of the ACHIEVE GREATER (Addressing Cardiometabolic Health In Populations Through Early PreVEntion in the GREAT LakEs Region) Center (IRB# 100221MP2A), the purpose of which is to improve cardiometabolic health in two uniquely comparable cities: Detroit, Michigan, and Cleveland, Ohio. The ACHIEVE GREATER Center involves separate but related projects that aim to improve cardiometabolic health outcomes through better risk factor control for three chronic conditions that are of tremendous public health importance, (hypertension (HTN), heart failure, and coronary heart disease), all of which contribute significantly to premature death in Detroit and Cleveland.

The present study is the prospective observational cohort component of ACHIEVE P1- EPI (Project 1) of the ACHIEVE GREATER Center and serves to characterize the population of patients with blood pressure (BP) levels above normal attending The Wayne Health Mobile Health Unit (MHU) events to better understand key factors (e.g., social determinants of health) that convey information about baseline BP levels and related clinical outcomes (e.g., follow-up clinic visits, BP control, and cardiovascular events).

DETAILED DESCRIPTION:
ACHIEVE P1- EPI aligns with the over-arching theme of the ACHIEVE GREATER center to reduce the burden of chronic cardiovascular disease in the urban Great Lakes region. It focuses on understanding key factors that drive the high prevalence and poor control of hypertension (HTN) in communities across metro Detroit. Much of this risk traces to social vulnerability and pervasive negative social determinants of health (SDoH) which impact access and quality of care. ACHIEVE P1- EPI is comprised of two main components: 1) a retrospective analysis of all MHU patients starting in April 2020 (IRB-23-04-5726); and 2) development of a prospective observational sub-cohort of MHU patients that consent to on-going follow up of their health care utilization and outcomes, a subset of whom will also consent to receive a home BP monitor where utilization of the device will be monitored.

This project focuses on the prospective component (ACHIEVE P1- EPI: Prospective), to enable the study team to characterize critical risk factors and track associations with subsequent health outcomes to inform a comprehensive preventative strategy to lower blood pressure (BP) and improve the control of early-stage HTN in the Detroit area.

ACHIEVE P1- EPI proposes an epidemiological approach to characterize key factors that convey information about baseline BP levels and/or that drive subsequent health outcomes. Using a combination of retrospective and prospective observational analytical approaches, the study team will leverage the Wayne Health Mobile Health Unit (MHU) platform to implement an observational cohort study that will characterize the antecedents, correlates and sequelae of abnormal blood pressure. The investigator and study team will also perform a nested randomized trial to determine if text message prompts improve the amount or quality of data collected remotely.

Key issues requiring elucidation are: the prevalence and predictors of negative SDoH among patients as well as their associations with screening BP levels and trajectories; the role of SDoH (and other factors) in determining the progression/remission of high BP over the following year; the rates and predictors of successful linkages with follow-up medical visits and receiving social services; the rates and predictors of the initiation of BP-lowering medications in subsequent clinical care; the persistence and predictors of follow-up clinical visits and treatments; the barriers and facilitators of linkages into the healthcare system; and the ultimate success rates and predictors of reaching BP goals. Answers to these questions will provide invaluable information to help guide data-driven improvements to the MHU program moving forward and inform future scalability in other regions and locations. These results will assist us in the optimizing and up-scaling of the program, including the development of improved strategies to successfully link individuals to social services and follow-up healthcare. The findings will help enhance the study team's overall care delivery pathways with the goals of improved BP control and reduced cardiometabolic health inequities in Detroit and beyond.

The specific aims are:

AIM-1: To develop a prospective observational cohort to observe subsequent health outcomes (e.g., blood pressure levels, cardiometabolic risk factors, clinic visits, medications, cardiovascular events) following MHU participation using Wayne health EMR dataset for follow-up. The study team will assess baseline predictors (e.g., SDoH, medications, demographics) of subsequent health outcomes and plan to probe area- and person-level profiles as potential sources of variation in appropriately developed multilevel models.

AIM-2: To develop a nested randomized trial of a sub-cohort to test for differences in adherence to a blood pressure measurement protocol among an intervention group that receives text message reminders and controls who instead receive standard of care without text message reminders. We will also test for differences in blood pressure profiles and, secondarily, emergency department utilization at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Mobile Health Unit Patients with blood pressure above normal (≥120 systolic and/or ≥80 mmHg)
* Has a phone with the ability to receive text messages
* 18+ years old
* Consent to allow prospective follow-up including through EHR review

Exclusion Criteria:

* Non-mobile health unit patients
* MHU patients with systolic BP < 120 mmHg AND diastolic BP < 80 mmHg
* Pregnant Women
* Children less than 18 years old
* Individuals viewed by the investigative team as unable to understand and sign the informed consent form
* Currently enrolled in another on-going interventional trial initiated on the mobile health unit

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-06-11 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Measure Blood Pressure Protocol Fidelity | 12 Months
  Achieve a minimum of six (6) measurements of two (2) or more readings of systolic and diastolic blood pressures at baseline, Month 6 and Month 11 within a seven (7) day period.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Korzeniewski, PhD, Principal Investigator — Wayne State University
Locations (1):
- Wayne Health Mobile Units, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided